CLINICAL TRIAL: NCT00535665
Title: The Clinical Trial of Pandemic Influenza Vaccine (Whole-Virion， Inactivated, Adjuvanted) on Healthy Adults by Randomized and Double-Blind Design: a Phase II Study
Brief Title: Safety and Immunogenicity of an Inactivated Pandemic Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-PanFlu-2001
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-11

CONDITIONS: Pandemic Influenza; Prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1: 10 ug, 14 days (Experimental)
  Interventions: Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14)
- 2: 5 ug, 28 days (Experimental)
  Interventions: Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14)
- 3: 10 ug, 28 days (Experimental)
  Interventions: Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14)
- 4: 15 ug, 28days (Experimental)
  Interventions: Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14)

INTERVENTIONS:
Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14) — two-dose regimen with 14 days apart: 5 microgram per dose
  Arms: 1: 10 ug, 14 days
Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14) — two-dose regimen with 28 days apart: 5 microgram per dose
  Arms: 2: 5 ug, 28 days
Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14) — two-dose regimen with 28 days apart: 10 microgram per dose
  Arms: 3: 10 ug, 28 days
Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14) — two-dose regimen with 28 days apart: 15 microgram per dose
  Arms: 4: 15 ug, 28days

SUMMARY:
A single center, randomized and double-blind phase II clinical trial is to be conducted in adults to evaluate the safety and immunogenicity of an inactivated pandemic influenza vaccine (whole-virion, aluminium-adjuvanted).

DETAILED DESCRIPTION:
The vaccine to be investigated is producted in embryonated hen's eggs using an H5N1 reference strain NIBRG-14 which was prepared by NIBSC. The strain is a reassortant between A/Vietnam/1194/2004 and A/PR/8/34 by reverse genetics.

Total 400 volunteers aged from 18 to 60 years old are to be enrolled with 100 subjects in each group. The eligible volunteers will receive two doses vaccine of 5μg，10μg or 15μg haemagglutinin antigen. The schedule is day 0,14 or day 0,28. The subjects will donate their blood samples for the detection of HI antibody and microneutralization antibody. Local and systematic adverse reactions will be recorded during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-60 years old
* Be able to show legal identity card for the sake of recruitment
* Be able to understand and sign the informed consent.

Exclusion Criteria:

* Woman： Who breast-feeding or planning to become pregnant during the 56 days of study participation
* Any history of allergic reactions was allergic to any component of the vaccine, such as eggs or ovalbumin;
* Any history of severe adverse reactions to vaccines, such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
* Autoimmune disease or immunodeficiency
* Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
* Diabetes mellitus (type I or II), with the exception of gestational diabetes
* History of thyroidectomy or thyroid disease that required medication within the past 12 months
* Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years
* Hypertension that was not well controlled by medication or is more than 145/95 mmHg at enrollment
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
* Active malignancy or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of study
* Seizure disorder other than:

  1. Febrile seizures under the age of two years old,
  2. Seizures secondary to alcohol withdrawal more than 3 years ago, or
  3. A singular seizure not requiring treatment within the last 3 years
* Asplenia, functional asplenia or any condition resulting in the absence or removal o the spleen
* Guillain-Barre Syndrome
* Women subjects with positive urinary pregnancy test
* Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
* History of any blood products administration within 3 months before the dosing
* Administration of any other investigational research agents within 30 days before the dosing
* Administration of any live attenuated vaccine within 30 days before the dosing
* Administration of subunit or inactivated vaccines, e.g. pneumococcal vaccine, or allergy treatment with antigen injections, within 14 days before the dosing
* Be receiving anti-TB prophylaxis or therapy currently
* Axillary temperature >37.0 centigrade at the time of dosing
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 402 (Actual)
Dates: Start 2007-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
HI antibody and Neutralization antibody | 0,28,42,56

SECONDARY OUTCOMES:
adverse reactions | 0,28,42,56

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wu, Principal Investigator — Beijing Centers for Diseases Control and Prevention

REFERENCES:
- [Derived] Wu J, Fang HH, Chen JT, Zhou JC, Feng ZJ, Li CG, Qiu YZ, Liu Y, Lu M, Liu LY, Dong SS, Gao Q, Zhang XM, Wang N, Yin WD, Dong XP. Immunogenicity, safety, and cross-reactivity of an inactivated, adjuvanted, prototype pandemic influenza (H5N1) vaccine: a phase II, double-blind, randomized trial. Clin Infect Dis. 2009 Apr 15;48(8):1087-95. doi: 10.1086/597401. PMID 19281330